CLINICAL TRIAL: NCT06526481
Title: Nasoseptal Double Flap Versus Rescue Flap in Endoscopic Transsphenoidal Pituitary Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MD.22.11.721
Record Dates: First submitted 2024-07-18; First posted 2024-07-29 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-07

CONDITIONS: Pituitary Adenoma
Keywords: pituitary surgery; double nasoseptal flap; rescue nasoseptal flap; nasal morbidity; transsphenoidal pituitary surgery
MeSH Terms: conditions — Pituitary Neoplasms

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single blinded study, only the participant is blinded to the group he is going to be in.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Double nasoseptal flap (Experimental): Nasoseptal double flap group:
  -On one side full sized nasoseptal flap will be elevated and a smaller sized nasoseptal flap will be elevated on the other side.
  Interventions: Procedure: Endoscopic Transsphenoidal pituitary surgery : Double Nasoseptal Flap Technique
- Rescue nasoseptal flap (Experimental): Nasoseptal rescue flap group:
  - A horizontal incision will be performed in the nasal septum in a posterior to anterior direction starting from the sphenoid ostium to a point opposite anterior end of the middle turbinate ( approximately up to one half of septum).
  Interventions: Procedure: Endoscopic Transsphenoidal pituitary surgery : Rescue Flap Technique

INTERVENTIONS:
Procedure: Endoscopic Transsphenoidal pituitary surgery : Double Nasoseptal Flap Technique — Patients with with symptomatic pituitary macroadenoma and tumor size ≥ 2 cm will have transsphenoidal endoscopic excision of pituitary adenoma.
  -On one side full sized nasoseptal flap will be elevated and a smaller sized nasoseptal flap will be elevated on the other side.
  Arms: Double nasoseptal flap
Procedure: Endoscopic Transsphenoidal pituitary surgery : Rescue Flap Technique — Patients with with symptomatic pituitary macroadenoma and tumor size ≥ 2 cm will have transsphenoidal endoscopic excision of pituitary adenoma.
  - A horizontal incision will be performed in the nasal septum in a posterior to anterior direction starting from the sphenoid ostium to a point opposite anterior end of the middle turbinate ( approximately up to one half of septum).
  Arms: Rescue nasoseptal flap

SUMMARY:
This paper investigates the outcomes of two surgical techniques-nasoseptal double flap and nasoseptal rescue flap-used in endoscopic transsphenoidal surgery for pituitary tumors. The nasoseptal flap technique has significantly reduced the incidence of postoperative Cerebrospinal Fluid (CSF) leaks but can cause nasal morbidity.

DETAILED DESCRIPTION:
The study aims to compare nasal morbidity and function between the two techniques in patients undergoing this type of surgery. Each patient's nasal morbidity, olfaction, and postoperative complications will be assessed using various tools.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients with symptomatic pituitary macroadenoma
* Tumor size ≥ 2 cm

Exclusion Criteria:

* -Absent sphenoid pneumatization.
* Temporal or frontal extension.
* Recurrent pituitary tumor after previous surgery.
* Previous nasal surgery.
* Associated nasal disease e.g. rhinosinusitis.
* Unfit for general anesthesia.
* Refusal of surgical intervention or signing consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2024-03-26 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Nasal morbidity | at baseline preoperative and 1 month and 3 months postoperative.
  Sinonasal Outcome Test 22 (SNOT-22) arabic translation questionnaire for nasal morbidity SinoNasal Outcome Test - 22 abbreviated (SNOT-22) includes 22 items for assessment by the patient. Each item is graded from 0 to 5. The minimum score is 0. The maximum score is 110. High score means higher nasal morbidity. Low scores mean better nasal morbidity.

SECONDARY OUTCOMES:
Operative data | at time of surgery
  Operative time

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad M. Al-Arman, Principal Investigator — Mansoura Faculty of Medicine, Masnoura University
Locations (1):
- Mansoura University, Department of otorhinolaryngology, Al Mansurah, Egypt